CLINICAL TRIAL: NCT00345748
Title: A Phase II, Multi-center, Randomized, Double-Blind, Placebo Controlled, Dose Response Study to Evaluate the Safety and Efficacy of Two Different Doses of Abatacept (BMS-188667) Administered Intravenously to Japanese Subjects With Active Rheumatoid Arthritis While Receiving Methotrexate
Brief Title: A Study of Abatacept in Japanese Patients With Active Rheumatoid Arthritis While Receiving Methotrexate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM101-071
Record Dates: First submitted 2006-06-23; First posted 2006-06-28 (Estimated); Last update posted 2011-04-25 (Estimated); Status verified 2011-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Abatacept 2 mg/kg (Active Comparator)
  Interventions: Drug: Abatacept
- Abatacept 10 mg/kg (Active Comparator)
  Interventions: Drug: Abatacept
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Abatacept — Injection, IV Infusion, Day 1, 15, 29 and every 28 days for 24 weeks
  Other Names: Orencia
  Arms: Abatacept 10 mg/kg; Abatacept 2 mg/kg
Drug: Placebo — Injectio, IV Infusion, Day 1, 15, 29 and every 28 days for 24 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to demonstrate that Abatacept combined with Methotrexate will demonstrate a dose response efficacy in Japanese subjects with active Rheumatoid Arthritis similar to the dose response efficacy previously observed in the International clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* patients with active Rheumatoid Arthritis while on methotrexate having 12 tender and 10 swollen joints at randomization

Exclusion Criteria:

* no current infection or other evolutive or uncontrolled disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2006-06; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Efficacy will be evaluated using the American College of Rheumatology response rate or ACR 20. This means the respective proportion of patients reaching an improvement of at least 20% of the ACR composite index from baseline. | at 6 months

SECONDARY OUTCOMES:
ACR 50 and ACR 70 will be assessed as respectively 50 and 70% improvement of the ACR composite index, quality of life by using SF36 questionnaire, Population Pharmacokinetics, Biomarkers, Immunogenicity | at 6 months
Safety (Severity of adverse events, causal relationship to the study drug, outcome, action taken with respect to the investigational product, treatment required) | at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (30):
- Japan (30):
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Goshogawara-Shi, Aomori
  - Local Institution, Chiba, Chiba
  - Local Institution, Fukui-shi, Fukui
  - Local Institution, Fukuoka, Fukuoka
  - Local Institution, Kitakyushu-Shi, Fukuoka
  - Local Institution, Higashi-Hiroshima-Shi, Hiroshima
  - Local Institution, Sapporo, Hokkaido
  - Local Institution, Kanzaki-Gun, Hyōgo
  - Local Institution, Kato-Gun, Hyōgo
  - Local Institution, Hitachi-Shi, Ibaraki
  - Local Institution, Tsukuba, Ibaraki
  - Local Institution, Sagamihara-Shi, Kanagawa
  - Local Institution, Sendai, Miyagi
  - Local Institution, Nagano, Nagano
  - Local Institution, Tsukubo-Gun, Okayama-ken
  - Local Institution, Kawachinagano-Shi, Osaka
  - Local Institution, Ureshino-Shi, Saga-ken
  - Local Institution, Iruma-Gun, Saitama
  - Local Institution, Kawagoe-Shi, Saitama
  - Local Institution, Kitamoto-Shi, Saitama
  - Local Institution, Hamamatsu, Shizuoka
  - Local Institution, Kawachigun, Tochigi
  - Local Institution, Tochigi, Tochigi
  - Local Institution, Arakawa-Ku, Tokyo
  - Local Institution, Bunkyo-Ku, Tokyo
  - Local Institution, Setagaya-Ku, Tokyo
  - Local Institution, Shinjuku-Ku, Tokyo
  - Local Institution, Takaoka-Shi, Toyama
  - Local Institution, Chiba